CLINICAL TRIAL: NCT03134404
Title: A Pilot Project to Assess the Feasibility of Integrating a Multidisciplinary Rapid Access Metastatic Bone Disease Program (RAMP) at The Ottawa Hospital
Brief Title: Project to Assess Feasibility of a Rapid Access Metastatic Bone Disease Program
Acronym: RAMP
Status: Withdrawn | Type: Observational
Why Stopped: study did not start
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: FORM ID 6174
Record Dates: First submitted 2016-12-21; First posted 2017-05-01 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Metastases to Bone
Keywords: RAMP; Rapid Access; Metastasis to Bone; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No Intervention — No Intervention is required for this study

SUMMARY:
The skeletal system is one of the most common sites for metastatic spread of many malignancies. Metastatic bone disease (MBD) can be associated with a significant reduction in quality of life due to debilitating pain and pathologic fractures. Multiple providers are involved in treating patients with MBD which can result in fragmented and delayed delivery of care. This fragmentation also leads to poor outcomes and patient experience. This project will assess whether it is feasible to integrate a multidisciplinary Rapid Access Metastatic Bone Disease Program (RAMP) at the Investigator's institution to improve the delivery of care to patients presenting with pelvic and lower extremity MBD. The goals of RAMP are: 1) Improve outcome and quality of care provided to MBD patients. 2) Improve patients experience through the participant's treatment journey. 3) Avert extra health care costs caused by unplanned admissions through ER and decrease redundancies due to unnecessary multiple clinic visits and double-ordering of diagnostic tests. This project will be designed to optimize the use of existing clinic resources more efficiently. Cancer patients and their loved ones will be actively engaged in the design of this project to better achieve its goals.

DETAILED DESCRIPTION:
More than 140,000 new cases of cancer are diagnosed annually in Canada, with nearly half of which metastasize to bone. The skeletal system is one of the most common sites for metastatic spread of many visceral malignancies, especially cancers originating from breast, prostate, lung, thyroid and kidney. Hematologic malignancies, such as multiple myeloma and lymphoma, also primarily manifest with multiple aggressive lytic lesions in the bone. A Skeletal Related Event (SRE) is the term given when a metastatic lesion arises in bone. With advances in effective systemic treatment and supportive care, the duration of survival of patients with bone metastases has improved substantially. This improvement in survival can be accompanied by significant morbidity and reduction in quality of life secondary to pain, pathologic fracture, and spinal cord compression from SREs. Pain and impaired mobility occur in approximately 65%-75% of patients with bone metastases. SREs are also associated with high economic burden secondary to increased costs of treatment and high rates of hospitalizations. It is estimated that a single episode of SRE can cost the medical system 36,462 USD. The current literature reflects significant diversity in the approach of diagnosing and treating MBD. Therefore, numerous studies have advocated the need for a multidisciplinary clinic to co-ordinate the diagnosis, treatment, and rehabilitation of patients with MBD patients. This strategy has also been proposed to improve the delivery of early and multimodal palliative management for patients in a cost effective approach.

Aims and Objectives: The aims of this project are: 1) Assess feasibility of establishing and integrating a multidisciplinary Rapid Access Metastatic Bone Disease Program (RAMP) at the Investigator's institution to improve the delivery of care to patients presenting with pelvic and lower extremity MBD. 2) Centralize referrals and streamline clinical care pathways for patients diagnosed with MBD to pelvis and lower extremity. 3) Assess improvement in outcome and patient experience. The objectives of this project are: 1) Establish a core multidisciplinary RAMP team to develop a patient-centered clinical care pathway for diagnosis and treatment. 2) Establish a standardized and rapid referral process for RAMP. 3) Triage consults and coordinate their integration into pre-existing weekly "musculoskeletal oncology" clinic at the cancer center. 4) Develop a centralized registry for patients presenting to RAMP to assess provider performance and evaluate the success of established clinical care pathways.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older and able to provide informed consent.
* Patient with an established tissue diagnosis of cancer.
* Patient with diagnosis of metastatic bone lesion which requires a referral to an Orthopedic Oncology Specialist.
* Patient will receive their care and treatment for this metastatic disease at The Ottawa Hospital.

Exclusion Criteria:

* Patient does not speak or understand adequate French or English to complete the functional outcome questionnaires.
* Patient has a documented cognitive impairment precluding questionnaire completion (e.g. dementia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are referred and subsequently followed for a diagnosis of Bone Metastatic Disease of the pelvis or lower extremities arising from a Primary Cancer elsewhere.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Standardization of the referral pathways | 2 years
  Identifying the rate of compliance from the ER, oncology (Medical, radiation and hematology), as well as primary physicians in directing referrals to RAMP. The goal is a compliance rate of 80%. This will be measured by capturing the consults for MBD of the pelvis and lower extremity that were referred outside RAMP referral pathway.

SECONDARY OUTCOMES:
Feasibility to triage MBD patients in currently existing musculoskeletal oncology clinics | 2 years
  The admission rate and triage of the musculoskeletal oncology clinic for MBD patients will help us identify the current systems true clinic capacity.
Improve patient flow and timely access to care. | 2 years
  This benefit will be measured by achieving wait time < 7 days for patients to be assessed for a pending pathologic fracture. The wait time will be captured by the RAMP registry which will keep meticulous track of all referral, visits and treatment dates.
Improvement in symptom management and patient satisfaction | 2 years
  This data will be captured by patients filling validated ESAS and patient.This data will be captured by patients filling validated ESAS and patient satisfaction questionnaires. These questionnaires will be collected during phase I (planning) of this project, and will be compared to surveys obtained during phase II(execution). We anticipate an improvement in patient satisfaction.

OTHER OUTCOMES:
Improvement in counseling MBD patients about mobility aids and fall risk assessment. | 2 years
  This metric can be captured by collaborating with our electronic chart experts (MOSAIQ) to create a field for RNs to document this item, which can then be tracked.

CONTACTS AND LOCATIONS:
Overall Officials: Hesham Abdelbary, MD, Principal Investigator — OHRI

IPD SHARING:
Plan to Share IPD: No